CLINICAL TRIAL: NCT00998686
Title: A Phase 3, Randomized, Double-Blind, Active-Controlled, Multi-Center Extension Study to Evaluate Safety and Efficacy of Dutogliptin in Subjects With Type 2 Diabetes Mellitus on a Background Medication of Metformin
Brief Title: Safety and Efficacy Study of Dutogliptin in Subjects With Type 2 Diabetes Mellitus on a Background Medication of Metformin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Phenomix (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Michael Huang, MD, Phenomix
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHX1149-PROT402
Record Dates: First submitted 2009-10-16; First posted 2009-10-20 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; DPP4 inhibitor; dutogliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dutogliptin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dutogliptin/PHX1149T (Experimental)
  Interventions: Drug: dutogliptin
- sitagliptin (Active Comparator)
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: dutogliptin — 400 mg
  Arms: dutogliptin/PHX1149T
Drug: sitagliptin — 100 mg
  Arms: sitagliptin

SUMMARY:
The purpose of this study is to demonstrate the safety and tolerability of dutogliptin over 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Completion of all required visits of a qualifying Phase 3 core protocol
* Current treatment of Type 2 diabetes mellitus as in PHX1149-PROT302

Exclusion Criteria:

* Any condition, disease, disorder or clinically relevant laboratory abnormality which, in the opinion of the investigator, would jeopardize the patient's appropriate participation in this study or obscure the effects of treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-10 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
To demonstrate safety and tolerability of dutogliptin as assessed by vital signs, adverse event reporting, routine clinical laboratory assessments, and ECG | 52 weeks

SECONDARY OUTCOMES:
To demonstrate maintenance or lowering of HbA1c and fasting plasma glucose | 52 weeks

CONTACTS AND LOCATIONS:
Locations (44):
- United States (23):
  - Phenomix Investigational Site 105, Montgomery, Alabama
  - Phenomix Investigational Site 121, Tempe, Arizona
  - Phenomix Investigational Site 137, Tempe, Arizona
  - Phenomix Investigational Site 105, Anaheim, California
  - Phenomix Investigational Site 103, Long Beach, California
  - Phenomix Investigational Site 106, Los Angeles, California
  - Phenomix Investigational Site 143, Coral Gables, Florida
  - Phenomix Investigational Site 142, Hialeah, Florida
  - Phenomix Investigational Site 133, Kissimmee, Florida
  - Phenomix Investigational Site 101, Honolulu, Hawaii
  - Phenomix Investigational Site 135, Chicago, Illinois
  - Phenomix Investigational Site 124, Indianapolis, Indiana
  - Phenomix Investigational Site 136, Brockton, Massachusetts
  - Phenomix Investigational Site 138, Biloxi, Mississippi
  - Phenomix Investigational Site 122, Las Vegas, Nevada
  - Phenomix Investigational Site 140, Las Vegas, Nevada
  - Phenomix Investigational Site 110, Trenton, New Jersey
  - Phenomix Investigational Site 116, Albuquerque, New Mexico
  - Phenomix Investigational Site 107, Winston-Salem, North Carolina
  - Phenomix Investigational Site 112, Greenville, South Carolina
  - Phenomix Investigational Site 102, Dallas, Texas
  - Phenomix Investigational Site 104, San Antonio, Texas
  - Phenomix Investigational Site 100, Kenosha, Wisconsin
- Argentina (3):
  - Phenomix Investigational Site 402, Buenos Aires
  - Phenomix Investigational Site 408, Buenos Aires
  - Phenomix Investigational Site 410, Mendoza
- Czechia (3):
  - Phenomix Investigational Site 208, Prague
  - Phenomix Investigational Site 209, Praha 4 Chodov
  - Phenomix Investigational Site 207, Uničov
- India (5):
  - Phenomix Investigational Site 707, Shāstrinagar, Jaipur
  - Phenomix Investigational Site 701, Bangalore, Karnataka
  - Phenomix Investigational Site 705, Trivandrum, Kerala
  - Phenomix Investigational Site 706, Indore, Madhya Pradesh
  - Phenomix Investigational Site 711, Mumbai, Maharashtra
- Peru (4):
  - Phenomix Investigational Site 607, Arequipa
  - Phenomix Investigational Site 601, Ica
  - Phenomix Investigational Site 604, Lima
  - Phenomix Investigational Site 610, Lima
- Poland (6):
  - Phenomix Investigational Site 300, Gdansk
  - Phenomix Investigational Site 309, Karkow
  - Phenomix Investigational Site 303, Katowice
  - Phenomix Investigational Site 306, Puławy
  - Phenomix Investigational Site 305, Warsaw
  - Phenomix Investigational Site 302, Wroclaw